CLINICAL TRIAL: NCT06947148
Title: The Impact of Comprehensive Post Hospital Management Based on Digital Health Intervention on Cardiac Function in Patients With Heart Failure: a Prospective, Multicenter, Randomized Controlled Study
Brief Title: The Impact of Comprehensive Post Hospital Management Based on DHI on Cardiac Function in Patients With HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yu Bo, Chief Physician, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KY2024-024
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure
Keywords: Heart Failure; Digital Health Intervention; Remote Dielectric Sensing; ReDS™; Comprehensive Health Care; 6 Min Walk Test; Randomized Controlled Trial
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive post hospital management group (Other): Based on the routine HF management of standard of care (SOC), the intervention group will carry out comprehensive post hospital management based on DHI, including cognitive behavioral therapy, digital self-monitoring and ReDS™ technology, etc.
  Interventions: Other: Comprehensive post hospital management based on digital health intervention(DHI)
- Routine Management Group (No Intervention): The routine management group will accept the routine HF management of SOC throughout the course, and the doctor will carry out treatment and management according to the actual clinical situation, including pre discharge education, precautions for commonly used drugs, guidance for daily life activities, etc.

INTERVENTIONS:
Other: Comprehensive post hospital management based on digital health intervention(DHI) — Based on the routine HF management of standard of care (SOC), the intervention group will carry out comprehensive post hospital management based on DHI, including cognitive behavioral therapy, digital self-monitoring and ReDS™ technology, etc.
  Arms: Comprehensive post hospital management group

SUMMARY:
Due to the complex nature of HF patients' conditions, long-term treatment and management are required, especially post hospital management, which is of great significance for improving patients' cardiac function and quality of life. With the increasing popularity of smartphones and the continuous development of medical technology, digital health intervention (DHI) has emerged as a new medical model in the treatment of diseases.

This study will establish a comprehensive post hospital management model of HF based on DHI, including cognitive behavioral therapy, digital self-monitoring and remote dielectric sensing (ReDS™) technology, etc., comprehensively strengthen the post hospital intervention and management of HF. Objective to explore the effect of comprehensive post hospital management based on DHI on cardiac function of patients with HF 6 months after discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized for HF, NYHA classification II-IV upon admission
2. The patient's residence is within the urban area of each center, and ReDS™ technology can be performed at home or at the outpatient clinic
3. No difficulty using smartphones, with basic Chinese reading and writing skills
4. Accept the terms and conditions of the study and obtain informed consent from the subjects/their families

Exclusion Criteria:

1. Age<21 years old
2. Patients with height<155 cm or>190 cm, BMI<22 kg/m2 or>36 kg/m2, chest circumference<80 cm or>115 cm, and flail chest or rib fractures
3. History of pulmonary embolism
4. chronic renal failure（Scr > 443umol/L）
5. History of heart transplantation or pacemaker implantation
6. Severe pulmonary hypertension
7. Suffering from end-stage chronic obstructive pulmonary disease, requiring home oxygen therapy
8. Massive pleural effusion
9. The subject is unable to complete the 6-minute walking test
10. Expected lifespan<6 months
11. Researchers believe that participants are not suitable to participate in this trial (such as pregnancy, severe visual or hearing impairment, etc.)
12. Individuals who are unable to understand and/or comply with this research procedure (such as those who are addicted to alcohol, substance abuse, or have mental illnesses)
13. Currently participating in clinical trials of other devices or drugs
14. Researchers involved in the design and execution of this study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | The 6th month after discharge
  Improvement in 6-minute walk test after discharge for 6 months

SECONDARY OUTCOMES:
Quality of life index (QLI) rating | The 1st ,3rd and 6th months after discharge
Kansas city cardiomyopathy questionnaire (KCCQ-23) rating | The 1st ,3rd and 6th months after discharge
NYHA classification | The 1st ,3rd and 6th months after discharge
Left ventricular ejection fraction (LVEF) | The 6th month after discharge
  Measured by echocardiography
Number of readmissions for heart failure | Within 6 months after discharge
  Number of readmissions for hospitalized patients with heart failure due to worsening heart failure after discharge
All-cause mortality | Within 6 months after discharge
Cardiac death | Within 6 months after discharge
  Any death caused by heart disease (such as myocardial infarction, low output HF, fatal arrhythmia), death without witnesses, death from unknown causes, and all surgery related deaths, including those related to concurrent treatment, are classified as cardiac death
Composite endpoint of all-cause death or readmission due to heart failure | Within 6 months after discharge
Time to first hospitalization for heart failure from baseline | Within 6 months after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China